CLINICAL TRIAL: NCT01015469
Title: International, Multi Centre, Open, Prospective, Randomized Study: Banded Versus Conventional Laparoscopic Roux-en-Y (GABY)
Brief Title: Banded Versus Conventional Laparoscopic Roux-en-Y (GABY)
Acronym: GABY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ClinTrio Ltd. (Other)
Responsible Party: Burkhart Frankenberger - Director-, ClinTrio Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IT5448081; EudraCT-No. 2009-016718-26
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Morbid Obesity Requiring Bariatric Surgery
Keywords: bariatric; surgery; obesity; Roux-en-Y; gastric; medical device; bypass; adiposity; GaBP-Ring; BMI; banded; laparoscopic
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Conventional laparoscopic Roux-en-Y gastric bypass (Golden Standard)
  Interventions: Procedure: Conventional laparoscopic Roux-en-Y gastric bypass
- Group B (Experimental): Conventional laparoscopic Roux-en-Y gastric bypass with additional restrictive silastic ring
  Interventions: Procedure: conventional laparoscopic Roux-en-Y gastric bypass with additional restrictive silastic ring

INTERVENTIONS:
Procedure: Conventional laparoscopic Roux-en-Y gastric bypass — Conventional laparoscopic Roux-en-Y gastric bypass
  Arms: Group A
Procedure: conventional laparoscopic Roux-en-Y gastric bypass with additional restrictive silastic ring — conventional laparoscopic Roux-en-Y gastric bypass with additional restrictive silastic ring (GaBP-Ring)
  Arms: Group B

SUMMARY:
Banded Versus Conventional Laparoscopic Roux-en-Y Gastric Bypass (GABY).

The aim of this novel study is to evaluate, if an additional restrictive silastic ring can avoid dilation of the gastro-entero anastomosis and adjacent small bowel with consecutive better postoperative weight loss and significantly improved long-term weight maintenance.

The study will not investigate the GaBP-Ring as medical product but the effect of the GaBP-Ring on weight loss in comparison to gastric bypass alone.

DETAILED DESCRIPTION:
GABY is designed as an international, multi center, open, prospective, randomized study to compare two methods of bariatric surgery: Banded versus conventional laparoscopic Roux-en-Y gastric bypass.

At least 16 international high volume centres of excellence in bariatric surgery and at least 384 patients (24 patients at each center) in total will be included into this study. At least 320 patients must have completed the study after 5 years.

Surgery will be performed according to standardized operating protocol. The group A (control group) will follow the worldwide golden standard of bariatric surgery (gastric bypass). Patients randomised to group B will receive in addition a restrictive silastic ring. The ring is a launched medical product and is registered in the European Community.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 40 kg /m2 to ≤ 50 kg/m2
* Eating habit: sweet eater and volume eater
* Signed informed consent
* Patients with one or more of the following comorbidities: Hypertension, Diabetes mellitus Type 2, Hyperlipidemia, Hyperuricemia, Sleep apnea, Degenerative diseases of: Spine osteochondrosis, hip, knee, feet

Exclusion Criteria:

* History of obesity surgery
* History of major abdominal surgery with consecutive malabsorption (no resections of the stomach, small and large bowel (exception: appendectomy)
* Patients not eligible to implement silastic ring size 6.5 cm
* History of drug or alcohol abuse
* History of major psychiatric illness conflicting with patient's compliance
* History of recent or chronic steroid medication
* Autoimmune disease
* Inflammatory bowel disease or malabsorptive disease
* Liver cirrhosis (CHILD B + C)
* Active viral or bacterial disease (e.g. HIV, Hepatitis B or C, Tbc etc.)
* Pregnant women or women with childbearing potential without efficient contraception
* History of cancer in the last five years
* Need of long-term anticoagulant medication for any reason
* Any medication with ingredient ASA

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Estimated)
Dates: Start 2009-02; Primary Completion 2014-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
postoperative reduction of body mass index (BMI) and maintenance related to used bariatric procedure | 0, 3, 6, 12 months and 2, 3, 4, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Konrad W Karcz, MD, Principal Investigator — Albert-Ludwigs-University of Freiburg
Locations (14):
- Hospital Hallein (Scientific Review Board), Hallein, Austria
- Belgium (3):
  - Hospital AZ St.-Jan AV, Bruges
  - AZ Sint-Blasius, Dendermonde
  - AZ Nikolaas, Sint-Niklaas
- Germany (5):
  - Privatpraxis Chirurgie bei Schlossparkklinik, Berlin
  - Albert-Ludwigs-University, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Chirurgische Klinik München-Bogenhausen GmbH, München
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
- Atruim Medical Centre, Heerlen, Netherlands
- Medical University of Lodz, Lodz, Poland
- Portugal (2):
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Hospital de Sao Sebastiano, Santa Maria de Feira
- International Medical Center, Jeddah, Saudi Arabia